CLINICAL TRIAL: NCT04165395
Title: A Randomized Controlled Trial of the Effectiveness of a Five-layer Foam Dressing and the Heelmedix Boot for the Acute Prevention of Sacral and Heel Pressure Ulcers After Spinal Cord Injury
Brief Title: Evaluate the Incidence of Sacral and Heel Pressure Ulcers During Acute Care After SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Medline Industries (Industry)
Responsible Party: Principal Investigator, Andréane Richard-Denis, Principal Investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-1636; ISS-2018-DIV31-014 (Other: Medline Industries, Inc.)
Record Dates: First submitted 2019-09-06; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-09

CONDITIONS: Spinal Cord Injuries
Keywords: Pressure Ulcers; Pressure Injury; Spinal Cord Injury; Prophylactic; Dressing
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Computer generated set of random numbers to determine group allocation with a ratio of 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will receive the standard of care adopted at Hôpital du Sacré-Coeur de Montréal in terms of pressure ulcers prevention in the SCI population.
- Intervention group (Experimental): In addition to undergoing the identical standard-of-care as the control group, all patients in this group will receive a prophylactic five-layer foam dressing placed directly on the sacral area and a Heelmedix boot installed alternately on both legs
  Interventions: Device: Five-layer foam dressing; Device: Heelmedix boot

INTERVENTIONS:
Device: Five-layer foam dressing — Five-layer foam dressing applied on the sacrum within 48 hours of spinal surgery
  Other Names: Opitfoam Gentle Silicone Faced Foam & Border Sacral Wound Dressing; MSC2377EP
  Arms: Intervention group
Device: Heelmedix boot — Heelmedix boot will be installed alternately from one foot to the other.
  Other Names: Heelmedix; MDT823330P, MDT823330SW, MDT823330XL
  Arms: Intervention group

SUMMARY:
This study evaluates the effect of the application of a five-layer foam dressing on the sacrum as well as a boot applied on the heels as preventive measures in the development of pressure ulcers in patients hospitalized with spinal cord injury. In order to study their effectiveness in preventing wounds, we will compare the number of wounds that developed on the sacrum and heels in participants with and without preventive treatments. The study will also assess the severity of pressure ulcers in participants with and without preventive treatment if they do develop. Half of the participants will receive the usual standard care for the prevention of pressure ulcers without dressing and boot, while the other half, in additon to standard of care, will also have a preventive dressing on the sacrum as well as Heelmedix boot applied alternately on each foot.

DETAILED DESCRIPTION:
Among all patient populations, individuals with spinaI cord injury are most vulnerable to pressure ulcers due to prolonged and severe immobilization, moisture exposure related to sphincters incontinence, friction and shear forces associated with difficult transfers, as well as abnormal micro vascular blood flow secondary to a disrupted autonomic function below the level of injury. These factors contribute to ischemia of the skin and underlying tissues over bony prominences, which lead to increased risk of pressure ulcers. Most severe spinal cord injuries are associated with higher risk of developing pressure ulcers and presenting more severe pressure ulcers. The sacral area and heels are most at risk for pressure ulcers in the spinal cord injury population. Consequently, prevention of pressure ulcers during the acute care hospitalization is of utmost importance. Patients will be randomized to the intervention group (prophylactic placement of foam dressing over sacrum and placement of a Heelmedix boot) or the control group (no prophylactic foam dressing over sacrum and no Heelmedix boot). Both groups will receive the standard-of-care at the facility for the prevention of pressure ulcers. The standard care can include a regular evaluation of the skin, a nutritional evaluation, the management of incontinence, the use of a gel mattress, the use of a low air loss pressure-reliving mattress, the use of safe patient mobilization, weekly assessment by a physiatrist, a change of position every 2 hours, as well as occupational therapy and physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male of female age 18 years of older;
* Admitted to Hôpital du Sacré-Coeur de Montréal for a traumatic or non-traumatic spinal cord injury;
* Spinal cord injury is either: Motor-complete (AIS A-B) or motor-incomplete (AIS C);
* Neurological level of injury is between C0 and L2;
* Patient or interpreter is able to understand English or French and provide informed consent.

Exclusion Criteria:

* AIS D Incomplete spinal cord injury;
* Cauda equina syndrome or neurological level of injury below L2;
* Sacral or heel pressure ulcer present at admission;
* Presence of dermatological disease or systemic disease that might interfere with the outcome assessment (active dermatitis, urticarial, etc.);
* Skin allergy to any components or ingredients of the foam dressing;
* Any medical condition that would endanger a patient treated with the foam dressing;
* Patient who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Compare the incidence of pressure ulcers at the sacrum during the acute care hospitalization after a SCI between patients treated with prophylactic five-layer foam dressing at the sacrum area and vs. controls | During the acute care hospitalization, approx 6 weeks
  Incidence of new PU at the sacrum during the acute care hospitilization
Compare the incidence of PU at the heel during the acute care hospitalization after a SCI between patients with placement of a prophylactic Heelmedix boot and controls | During the acute care hospitalization, approx 6 weeks
  Incidence of new PU at the heel area during the acute care hospitilization

SECONDARY OUTCOMES:
Compare the severity of PU at the sacrum during the acute care hospitalization after a SCI between patients treated with prophylactic five-layer foam dressing at the sacrum area and controls | During the acute care hospitalization, approx 6 weeks
  Grade of PU based on the NPUAP grading system
Compare the severity of PU at the heel during the acute care hospitalization after a SCI between patients with placement of a prophylactic Heelmedix boot and controls | During the acute care hospitalization, approx 6 weeks
  Grade of PU based on the NPUAP grading system

CONTACTS AND LOCATIONS:
Overall Officials: Andréane Richard-Denis, M.D., MSC., Principal Investigator — CIUSSS du Nord-de-l'Île-de-Montréal-Hôpital du Sacré-Cœur de Montréal; Jean-Marc Mac-Thiong, M.D., Ph. D.,, Study Director — CIUSSS du Nord-de-l'Île-de-Montréal-Hôpital du Sacré-Cœur de Montréal
Locations (1):
- CIUSSS du Nord-de-l'Île-de-Montréal-Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denis AR, Feldman D, Thompson C, Mac-Thiong JM. Prediction of functional recovery six months following traumatic spinal cord injury during acute care hospitalization. J Spinal Cord Med. 2018 May;41(3):309-317. doi: 10.1080/10790268.2017.1279818. Epub 2017 Feb 15. PMID 28198660
- [Background] Thompson C, Mutch J, Parent S, Mac-Thiong JM. The changing demographics of traumatic spinal cord injury: An 11-year study of 831 patients. J Spinal Cord Med. 2015 Mar;38(2):214-23. doi: 10.1179/2045772314Y.0000000233. Epub 2014 Aug 6. PMID 25096709
- [Background] Richard-Denis A, Feldman DE, Thompson C, Mac-Thiong JM. The impact of acute management on the occurrence of medical complications during the specialized spinal cord injury acute hospitalization following motor-complete cervical spinal cord injury. J Spinal Cord Med. 2018 Jul;41(4):388-396. doi: 10.1080/10790268.2017.1350331. Epub 2017 Jul 19. PMID 28724333
- [Background] Richard-Denis A, Thompson C, Bourassa-Moreau E, Parent S, Mac-Thiong JM. Does the Acute Care Spinal Cord Injury Setting Predict the Occurrence of Pressure Ulcers at Arrival to Intensive Rehabilitation Centers? Am J Phys Med Rehabil. 2016 Apr;95(4):300-8. doi: 10.1097/PHM.0000000000000381. PMID 26418488
- [Background] Richard-Denis A, Beausejour M, Thompson C, Nguyen BH, Mac-Thiong JM. Early Predictors of Global Functional Outcome after Traumatic Spinal Cord Injury: A Systematic Review. J Neurotrauma. 2018 Aug 1;35(15):1705-1725. doi: 10.1089/neu.2017.5403. Epub 2018 Apr 17. PMID 29455634
- [Background] Padula WV, Mishra MK, Makic MB, Sullivan PW. Improving the quality of pressure ulcer care with prevention: a cost-effectiveness analysis. Med Care. 2011 Apr;49(4):385-92. doi: 10.1097/MLR.0b013e31820292b3. PMID 21368685
- [Background] Santamaria N, Gerdtz M, Sage S, McCann J, Freeman A, Vassiliou T, De Vincentis S, Ng AW, Manias E, Liu W, Knott J. A randomised controlled trial of the effectiveness of soft silicone multi-layered foam dressings in the prevention of sacral and heel pressure ulcers in trauma and critically ill patients: the border trial. Int Wound J. 2015 Jun;12(3):302-8. doi: 10.1111/iwj.12101. Epub 2013 May 27. PMID 23711244
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Background] Edsberg LE, Black JM, Goldberg M, McNichol L, Moore L, Sieggreen M. Revised National Pressure Ulcer Advisory Panel Pressure Injury Staging System: Revised Pressure Injury Staging System. J Wound Ostomy Continence Nurs. 2016 Nov/Dec;43(6):585-597. doi: 10.1097/WON.0000000000000281. PMID 27749790
- See also: Wound Source — http://www.woundsource.com/patientcondition/pressure-injuries-stage-1